CLINICAL TRIAL: NCT01642992
Title: Korean Coronary Bifurcation Stenting (COBIS) Registry II
Status: Completed | Type: Observational
Sponsor: Hyeon-Cheol Gwon (Other)
Responsible Party: Sponsor-Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2010-11-060
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Bifurcation Lesion
Keywords: Coronary bifurcation lesion; Drug-eluting stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Coronary bifurcation lesion

SUMMARY:
The COBIS II registry is a multi-center, real-world registry of drug-eluting stenting in coronary bifurcation lesions in South Korea. From 18 major coronary intervention centers in Korea, a total of 2,873 patients were enrolled in this database between January 2003 and December 2009.

The aim of the study was to investigate long-term clinical results and predictors of adverse outcomes after percutaneous coronary intervention with drug-eluting stents for coronary bifurcation lesions in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Any type of bifurcation lesion in major epicardial artery
* Side branch reference diameter >= 2.3 mm and at least stentable with 2.5 mm stent
* Treated with drug-eluting stent

Exclusion Criteria:

* Protected left main disease previous CABG for LAD or LCX territory
* Cardiogenic Shock
* History of CPR in the same hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary bifurcation lesion treated with drug-eluting stents
Sampling Method: Probability Sample
Enrollment: 2873 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of the composite outcomes of cardiac death, target vessel-related myocardial infarction, or target-lesion revascularization | 3 years

SECONDARY OUTCOMES:
Cardiac death | 3 years
Myocardial infarction | 3 years
Target lesion revascularization | 3 years
Stent thrombosis | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi KH, Bruno F, Cho YK, De Luca L, Song YB, Kang J, Mattesini A, Gwon HC, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Hur SH, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, D'Ascenzo F, Nam CW, de Filippo O. Comparison of Outcomes Between 1- and 2-Stent Techniques for Medina Classification 0.0.1 Coronary Bifurcation Lesions. JACC Cardiovasc Interv. 2023 Sep 11;16(17):2083-2093. doi: 10.1016/j.jcin.2023.06.013. Epub 2023 Aug 9. PMID 37565964
- [Derived] Lee JM, Lee SH, Kim J, Choi KH, Park TK, Yang JH, Song YB, Hahn JY, Choi JH, Choi SH, Kim HS, Chun WJ, Nam CW, Hur SH, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Lim DS, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Hong SJ, Koo BK, Gwon HC. Ten-Year Trends in Coronary Bifurcation Percutaneous Coronary Intervention: Prognostic Effects of Patient and Lesion Characteristics, Devices, and Techniques. J Am Heart Assoc. 2021 Sep 21;10(18):e021632. doi: 10.1161/JAHA.121.021632. Epub 2021 Sep 13. PMID 34514841
- [Derived] Yang JH, Lee JM, Park TK, Song YB, Hahn JY, Choi JH, Choi SH, Yu CW, Chun WJ, Oh JH, Koo BK, Jeong JO, Kim HS, Gwon HC. The Proximal Optimization Technique Improves Clinical Outcomes When Treated without Kissing Ballooning in Patients with a Bifurcation Lesion. Korean Circ J. 2019 Jun;49(6):485-494. doi: 10.4070/kcj.2018.0352. Epub 2019 Feb 22. PMID 30891962
- [Derived] Jang WJ, Ahn SG, Song YB, Choi SH, Chun WJ, Oh JH, Cho SW, Kim BS, Yoon JH, Koo BK, Yu CW, Jang YS, Tahk SJ, Kim HS, Gwon HC, Lee SY, Hahn JY. Benefit of Prolonged Dual Antiplatelet Therapy After Implantation of Drug-Eluting Stent for Coronary Bifurcation Lesions: Results From the Coronary Bifurcation Stenting Registry II. Circ Cardiovasc Interv. 2018 Jul;11(7):e005849. doi: 10.1161/CIRCINTERVENTIONS.117.005849. PMID 30006330
- [Derived] Yu CW, Yang JH, Song YB, Hahn JY, Choi SH, Choi JH, Lee HJ, Oh JH, Koo BK, Rha SW, Jeong JO, Jeong MH, Yoon JH, Jang Y, Tahk SJ, Kim HS, Gwon HC. Long-Term Clinical Outcomes of Final Kissing Ballooning in Coronary Bifurcation Lesions Treated With the 1-Stent Technique: Results From the COBIS II Registry (Korean Coronary Bifurcation Stenting Registry). JACC Cardiovasc Interv. 2015 Aug 24;8(10):1297-1307. doi: 10.1016/j.jcin.2015.04.015. PMID 26315732
- [Derived] Song YB, Hahn JY, Yang JH, Choi SH, Choi JH, Lee SH, Jeong MH, Kim HS, Lee JH, Yu CW, Rha SW, Jang Y, Yoon JH, Tahk SJ, Seung KB, Oh JH, Park JS, Gwon HC. Differential prognostic impact of treatment strategy among patients with left main versus non-left main bifurcation lesions undergoing percutaneous coronary intervention: results from the COBIS (Coronary Bifurcation Stenting) Registry II. JACC Cardiovasc Interv. 2014 Mar;7(3):255-63. doi: 10.1016/j.jcin.2013.11.009. Epub 2014 Feb 13. PMID 24529936
- [Derived] Hahn JY, Chun WJ, Kim JH, Song YB, Oh JH, Koo BK, Rha SW, Yu CW, Park JS, Jeong JO, Choi SH, Choi JH, Jeong MH, Yoon JH, Jang Y, Tahk SJ, Kim HS, Gwon HC. Predictors and outcomes of side branch occlusion after main vessel stenting in coronary bifurcation lesions: results from the COBIS II Registry (COronary BIfurcation Stenting). J Am Coll Cardiol. 2013 Oct 29;62(18):1654-1659. doi: 10.1016/j.jacc.2013.07.041. Epub 2013 Aug 14. PMID 23954335